CLINICAL TRIAL: NCT00740129
Title: An Open Label, Reclast®/Aclasta®, Re-treatment of Relapsed Patients With Paget's Disease of Bone Who Participated in the CZOL446K2304 and CZOL446K2305 Core Registration Studies
Brief Title: Re-treatment of Participants With Paget's Disease Using Zoledronic Acid
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CZOL446K2418; 2008-002898-12 (EudraCT Number)
Record Dates: First submitted 2008-08-21; First posted 2008-08-22 (Estimated); Results first posted 2021-05-26 (Actual); Last update posted 2021-05-26 (Actual); Status verified 2021-05

CONDITIONS: Paget's Disease of the Bone
Keywords: Paget's Disease; Zoledronic acid; Reclast®/Aclasta®; Infusion; Re-treatment; Re-lapse
MeSH Terms: conditions — Osteitis Deformans | interventions — Zoledronic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Zoledronic Acid 5 mg (Experimental): Participants received single re-treatment dose of zoledronic acid 5 mg intravenous (IV) infusion.
  Interventions: Drug: Zoledronic Acid

INTERVENTIONS:
Drug: Zoledronic Acid — Zoledronic acid 5 mg intravenous infusion once
  Other Names: Reclast®/Aclasta®

SUMMARY:
The purpose of this study was to demonstrate that participants with Paget's disease of the bone who had responded to zoledronic acid treatment as participants in the core registration studies CZOL446K2304 and CZOL446K2305 and later experienced a relapse can be successfully treated with a 5 milligram (mg) infusion of zoledronic acid.

DETAILED DESCRIPTION:
Uncontrolled study

ELIGIBILITY:
Inclusion Criteria:

* Written Informed Consent
* Participants with Paget's disease randomized to the zoledronic acid arm from the CZOL446K2304 and CZOL446K2305 core studies and who were responders by 6 months
* Confirmed relapse of Paget's disease of bone (i.e., serum alkaline phosphatase (SAP) above upper limit of normal (ULN), bone scan, worsening clinical symptoms)

Exclusion Criteria:

* A participant previously treated with zoledronic acid who relapsed and was retreated with anti-resorptive bisphosphonate or calcitonin therapy within the last 12 months
* Bisphosphonate Hypersensitivity
* Participants with suspected/proven metastases at re-treatment
* Calculated creatinine clearance <35 milliliter/minute (mL/min) at screening
* Serum calcium level <2.07 millimole/liter (mmol/L) at screening
* Active primary hyperparathyroidism, hyperparathyroidism, hypoparathyroidism or hypothyroidism

Other protocol-defined inclusion/exclusion criteria may apply.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2008-10-21 (Actual); Primary Completion 2011-03-14 (Actual); Study Completion 2011-03-14 (Actual)

CONTACTS AND LOCATIONS:
Locations (11):
- Novartis Investigative site, Brussels, Belgium
- Canada (2):
  - Novartis Investigative site, Montreal
  - Novartis Investigative site, Québec
- Novartis Investigative site, Auckland, New Zealand
- Novartis Investigative site, Cape Town, South Africa
- Spain (4):
  - Novartis Investigative site, Barcelona
  - Novartis Investigative site, Madrid
  - Novartis Investigative site, Salamanca
  - Novartis Investigative site, Valencia
- United Kingdom (2):
  - Novartis Investigative site, Nottingham
  - Novartis Investigative site, Oxford

REFERENCES:
- [Result] Reid IR, Brown JP, Levitt N, Roman Ivorra JA, Bachiller-Corral J, Ross IL, Su G, Antunez-Flores O, Aftring RP. Re-treatment of relapsed Paget's disease of bone with zoledronic acid: results from an open-label study. Bonekey Rep. 2013 Nov 6;2:442. doi: 10.1038/bonekey.2013.176. eCollection 2013. PMID 24422139

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 6 participants from core studies CZOL44K2304 and CZOL44K2305 who met the definition of responders at the end of study visit but later relapsed during the extension of observation period took part in the study at 5 investigative sites in Canada, Spain, New Zealand and, South Africa from 21 October 2008 to 14 March 2011.
Groups:
- Zoledronic Acid 5 mg: Participants received single re-treatment dose of zoledronic acid 5 mg IV infusion.
Period: Overall Study
Arm/Group | Zoledronic Acid 5 mg
Started | 6
Completed | 6
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Intent-to-Treat (ITT) Population included all enrolled participants who were previously randomized to zoledronic acid in the core studies (CZOL44K2304 and CZOL44K2305) and who received the intravenous study drug in this retreatment study.
Arm/Group | Zoledronic Acid 5 mg
Number analyzed (Participants) | 6
Age, Continuous [Mean (Standard Deviation); unit: years] | 75.2 (6.08)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 4
Baseline Serum Alkaline Phosphatase [Mean (Standard Deviation); unit: Units/Liter (U/L)] | 200.3 (59.62)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Serum Alkaline Phosphatase Within the Normal Range at Month 6 Last Observation Carried Forward (LOCF)
Description: Normalization of serum alkaline phosphatase (SAP) occurred if the SAP measurement fell within the normal ranges. The lower and upper limits of normal ranges were 31 and 110 Units/Liter (U/L) for participants with age ≤ 58 years old and 35 and 115 U/L for participants with age > 58 years old, respectively. Last observation carried forward (LOCF) was defined as the last post-baseline SAP value prior to month 6 for a participant who did not have an SAP value at month 6.
Time Frame: Month 6
Population: Modified Intent-to-Treat (MITT) Population included all enrolled participants who were previously randomized to zoledronic acid in the core studies (CZOL44K2304 and CZOL44K2305) and received the intravenous study drug and had baseline and at least one post-baseline assessment of the serum SAP in this retreatment study.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Zoledronic Acid 5 mg
Number analyzed (Participants) | 6
Percentage of Participants | 83.3 [35.9 to 99.6]

2. Secondary Outcome: Percentage Change From Baseline in Serum Alkaline Phosphatase (SAP) Levels
Description: The percentage change in SAP at Months 3 and 6 relative to baseline were measured.
Time Frame: Baseline, Months 3 and 6
Population: MITT Population included all enrolled participants who were previously randomized to zoledronic acid in the core studies (CZOL44K2304 and CZOL44K2305) and received the intravenous study drug and had baseline and at least one post-baseline assessment of the serum SAP in this retreatment study.
Measure: Mean (Standard Error); unit: percentage change
Arm/Group | Zoledronic Acid 5 mg
Number analyzed (Participants) | 6
percentage change
  Percentage Change From Baseline in SAP Level at Month 3 | -53.12 (7.607)
  Percentage Change From Baseline in SAP Level at Month 6 | -49.51 (10.090)

3. Secondary Outcome: Percentage of Participants With SAP Within the Normal Range
Description: Normalization of SAP occurred if the SAP measurement fell within the normal ranges. The lower and upper limits of normal ranges were 31 and 110 Units/Liter (U/L) for participants with age ≤ 58 years old and 35 and 115 U/L for participants with age > 58 years old, respectively.
Time Frame: Months 3 and 6
Population: MITT Population included all enrolled participants who were previously randomized to zoledronic acid in the core studies (CZOL44K2304and CZOL44K2305) and received the intravenous study drug and had baseline and at least one post-baseline assessment of the serum SAP in this retreatment study.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Zoledronic Acid 5 mg: Participants received single re-treatment dose of zoledronic acid 5 mg by IV infusion.
Arm/Group | Zoledronic Acid 5 mg
Number analyzed (Participants) | 6
percentage of participants
  Month 3 | 100.0 [54.1 to 100.0]
  Month 6 | 83.3 [35.9 to 99.6]

4. Secondary Outcome: Number of Participants With At Least One or More Treatment-Emergent Adverse Events (TEAEs)
Description: Adverse event was the appearance or worsening of any undesirable sign, symptom, or medical condition that occurred after starting the study drug even if the event was not considered to be related to study drug. TEAEs were defined as AEs that were absent prior to, but occurred after the i.v. infusion of study drug. TEAEs also included those that were present prior to the i.v. study drug infusion (i.e., as part of the extended observation period) but occurred at an increased severity after the i.v. infusion of study drug.
Time Frame: 6 months
Population: Safety Population included all enrolled participants previously randomized to zoledronic acid in the core studies (CZOL44K2304 and CZOL44K2305) who received intravenous study drug in this retreatment study.
Measure: Count of Participants; unit: Participants
Arm/Group | Zoledronic Acid 5 mg
Number analyzed (Participants) | 6
Participants | 1

5. Other Pre Specified Outcome: Collect Information Pertaining to Relapse Diagnosis to Define Retreatment Guidelines for Paget's Disease
Time Frame: 6 months
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Zoledronic Acid 5 mg
All-Cause Mortality (participants affected / at risk) | 0/6
Serious Adverse Events (participants affected / at risk) | 0/6
Other Adverse Events (participants affected / at risk) | 1/6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Zoledronic Acid 5 mg (N=6)
Influenza (Infections and infestations) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.